CLINICAL TRIAL: NCT05687916
Title: A Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of TAK-861 for the Treatment of Narcolepsy Without Cataplexy (Narcolepsy Type 2)
Brief Title: A Study of TAK-861 in Participants With Narcolepsy Type 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-861-2002; 2022-002966-34 (EudraCT Number); U1111-1282-8382 (Other: WHO Universal Trial Number); jRCT2031230050 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Narcolepsy Type 2
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo tablets matching TAK-861, orally, twice daily (BID), from Days 1 to 56.
  Interventions: Drug: Placebo
- TAK-861 2 milligrams (mg) BID (Experimental): Participants received TAK-861 2 mg, orally, BID, from Days 1 to 56.
  Interventions: Drug: TAK-861 2 mg
- TAK-861 2 mg and 5 mg (Experimental): Participants received TAK-861 2 mg followed by the 5 mg dose, orally, from Days 1 to 56.
  Interventions: Drug: TAK-861 2 mg and 5 mg

INTERVENTIONS:
Drug: Placebo — TAK-861 placebo matching tablets.
  Arms: Placebo
Drug: TAK-861 2 mg — TAK-861 2 mg tablets.
  Arms: TAK-861 2 milligrams (mg) BID
Drug: TAK-861 2 mg and 5 mg — TAK-861 2 mg and 5 mg tablets.
  Arms: TAK-861 2 mg and 5 mg

SUMMARY:
The main aim is to evaluate the effect of TAK-861 on symptoms of narcolepsy, including excessive daytime sleepiness (EDS) as measured by sleep latency from the Maintenance of Wakefulness Test (MWT).

The study will enroll approximately 60 participants and they will be randomly assigned to 3 groups (20 per group) to take one of two different doses of TAK-861 or a placebo. All the participants will receive the treatment for 8 weeks. Participants will be asked to complete some questionnaires during the study. This trial will be conducted in North America, Europe, and Asia Pacific.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-861. TAK-861 is being tested to treat people who have narcolepsy without cataplexy [Narcolepsy Type 2 (NT2)]. This study will evaluate the efficacy, safety, and tolerability of 2 oral doses of TAK-861.

The study will enroll approximately 60 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-861 Dose 1
* TAK-861 Dose 2
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

This is a multi-center trial to be conducted worldwide. The overall time to participate in this study is approximately 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

- The participant is aged 18 to 70 years, inclusive, at the time of signing the informed consent form (ICF).

Note: In Japan, participants aged 16 to 70 years, inclusive, may be included.

- The participant has an International Classification of Sleep Disorders, 3rd edition (ICSD-3) diagnosis of NT2 by preceding polysomnography (PSG)/ multiple sleep latency test (MSLT), performed within the past 5 years.

Note: If there is a potential participant with NT2 for whom a diagnostic nocturnal polysomnography (nPSG)/MSLT was performed more than 5 years ago or is not available, the site may repeat the diagnostic PSG/MSLT.

Exclusion Criteria:

* The participant has a current medical disorder, other than narcolepsy without cataplexy, associated with EDS.
* The participant has history of epilepsy, seizure, or convulsion, or has a family history of inherited disorders associated with seizure (except for a single febrile seizure in childhood).
* The participant has one or more of the following psychiatric disorders:

  1. Any current unstable psychiatric disorder.
  2. Current or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including schizoaffective disorder, major depression with psychotic features, bipolar depression with psychotic features, obsessive compulsive disorder, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
  3. Current diagnosis or history of substance use disorder as defined in the DSM-5. Note: If the history of substance use disorder is more than 12 months before baseline, the participant may be allowed to enroll in the study after consultation with the sponsor or designee. (Participant must also have negative urine drug screen at the screening and Day -2 visit.)
  4. Current active major depressive episode (MDE) or who have had an active MDE in the past 6 months.
* The participant has a history of cerebral ischemia, transient ischemic attack (<5 years ago), intracranial aneurysm, or arteriovenous malformation.
* The participant had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks before the screening visit.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (56):
- United States (22):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Mayo Clinic Arizona-PPDS, Scottsdale, Arizona
  - Stanford Center for Sleep Sciences and Medicine, Redwood City, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Delta Waves LLC - Hunt - PPDS, Colorado Springs, Colorado
  - Florida Pediatric Research Institute, Orlando, Florida
  - Neurotrials Research, Atlanta, Georgia
  - Georgia Neuro Center, Gainesville, Georgia
  - Neurocare Inc., Newton, Massachusetts
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - St. Lukes Sleep Medicine and Research Center, Chesterfield, Missouri
  - Research Carolina Elite, Denver, North Carolina
  - ARSM Research, LLC, Huntersville, North Carolina
  - Tricoastal Narcolepsy and Sleep Disorders Center, PLLC, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Comprehensive Sleep Medicine Associates - Sugar Land, Houston, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas
  - Children's Specialty Group, Norfolk, Virginia
- Woolcock Institute of Medical Research, Glebe, New South Wales, Australia
- Terveystalo Helsinki Sleep Clinic, Helsinki, Uusimaa, Finland
- France (3):
  - Hopital Saint-Eloi, Montpellier, Herault
  - CHU de Grenoble, La Tronche, Isere
  - Hopital de la Pitie Salpetriere, Paris
- Germany (2):
  - Somni Bene Institut fur Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Advanced Sleep Research GmbH, Berlin
- Italy (3):
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Istituto Neurologico Mediterraneo Neuromed, Pozzilli, Molise
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bellaria
- Japan (11):
  - Akita University Hospital, Akita, Akita
  - Ehime University Hospital, Toon-Shi, Ehime
  - You Ariyoshi Sleep Clinic, Kitakyushu, Hukuoka
  - Kurume University Hospital, Kurume-Shi, Hukuoka
  - Howakai Kuwamizu Hospital, Kumamoto, Kumamoto
  - Gokeikai Osaka Kaisei Hospital, Osaka, Osaka
  - Koishikawa Tokyo Hospital, Bunkyo-Ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira-Shi, Tokyo
  - Yoyogi Sleep Disorder Center, Shibuya-Ku, Tokyo
  - Aichi Medical University Hospital, Nagakute
  - RESM respiratory and sleep medical-care clinic, Yokohama
- Netherlands (2):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Slaap-Waakcentrum SEIN Heemstede, Heemstede, North Holland
- Oslo Universitetssykehus HF Rikshospitalet, Oslo, Norway
- Spain (6):
  - Hospital Universitario Araba Santiago, Vitoria-Gasteiz, Alava
  - Hospital General Universitari de Castello, Castellon, Castellon
  - Hospital de La Ribera, Alzira, Valencia
  - Hospital Clinic de Barcelona, Barcelona
  - Instituto de Investigaciones del Sueno, Madrid
  - Hospital Vithas Madrid Arturo Soria, Madrid
- Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County, Sweden
- Switzerland (3):
  - Klinik Barmelweid AG, Barmelweid, Aargau (de)
  - Neurocenter of Southern Switzerland, Lugano, Ticino (it)
  - Universitaetsspital Bern - Inselspital, Bern

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/b8004ec7e72e4dd0?idFilter=%5B%22TAK-861-2002%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 28 investigative sites globally from 09 January 2023 to 25 December 2023.
Pre-assignment Details: Participants with a diagnosis of narcolepsy type 2 (NT2) were enrolled in the study to receive either TAK-861 or placebo.
Groups:
- TAK-861 2 mg BID: Participants received TAK-861 2 milligrams (mg), orally, BID, from Days 1 to 56.
Period: Overall Study
Arm/Group | Placebo | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg
Started | 24 | 23 | 24
Completed | 21 | 19 | 22
Not Completed | 3 | 4 | 2
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Reason not Specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo tablets matching TAK-861, orally, BID, from Days 1 to 56.
- TAK-861 2 mg BID: Participants received TAK-861 2 mg, orally, BID, from Days 1 to 56.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg | Total
Number analyzed (Participants) | 24 | 23 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.69) | 34.9 (9.77) | 36.8 (12.61) | 36.2 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 17 | 49
  Male | 6 | 9 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 2 | 13
  Not Hispanic or Latino | 18 | 18 | 20 | 56
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 1 | 5 | 13
  White | 13 | 19 | 14 | 46
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Average Sleep Latency From the Maintenance of Wakefulness Test (MWT) [Mean (Standard Deviation); unit: minutes] — The MWT is a validated, objective measure that evaluates a participant's ability to remain awake under soporific conditions for a defined period. During each MWT session (1 session = 40 minutes), participants were instructed to sit quietly and remain awake for as long as possible. Sleep latency in each session was recorded on electroencephalography (EEG). If no sleep was observed according to these rules, then the latency was defined as 40 minutes.
  minutes | 10.8 (8.72) | 9.9 (10.29) | 8.4 (8.26) | 9.7 (9.04)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Sleep Latency as Determined From the MWT at Week 8
Description: The MWT is a validated, objective measure that evaluates a participant's ability to remain awake under soporific conditions for a defined period. During each MWT session (1 session = 40 minutes), participants were instructed to sit quietly and remain awake for as long as possible. Sleep latency in each session was recorded on EEG. If no sleep was observed according to these rules, then the latency was defined as 40 minutes. The linear mixed effects model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline, Week 8
Population: The Full Analysis Set included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 post-dose efficacy measurement. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg
Number analyzed (Participants) | 21 | 19 | 22
minutes | 2.14 (2.246) | 1.90 (2.384) | 4.54 (2.300)
Statistical Analysis 1: Comparison: Placebo vs TAK-861 2 mg BID; Test type: Superiority; p = 0.989, MMRM — The analysis used a linear MMRM with fixed effects for Baseline, age, prior use of narcolepsy medications, treatment, visit, and treatment-by-visit interaction as covariates. Reported p-value is adjusted for multiplicity; An unstructured variance-covariance structure was used; LS Mean Difference Estimate = -0.24, 95% CI 2-sided [-6.67 to 6.18], Standard Error of Mean 3.277
Statistical Analysis 2: Comparison: Placebo vs TAK-861 2 mg and 5 mg; Test type: Superiority; p = 0.916, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; LS Mean Difference Estimate = 2.4, 95% CI 2-sided [-3.93 to 8.72], Standard Error of Mean 3.227

2. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score at Week 8
Description: The ESS is a subjective, self-administered, validated scale (scored 0 to 3) to respond to each of the 8 questions of daily life that asks participants how likely they are to fall asleep in those situations. The scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range. The MMRM was used for analysis.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg
Number analyzed (Participants) | 20 | 19 | 22
score on a scale | -3.39 (1.140) | -3.71 (1.206) | -6.45 (1.121)
Statistical Analysis 1: Comparison: Placebo vs TAK-861 2 mg BID; Test type: Superiority; p = 0.989, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; LS Mean Difference Estimate = -0.32, 95% CI 2-sided [-3.57 to 2.92], Standard Error of Mean 1.656 — LS in LS Mean Difference denotes least squares
Statistical Analysis 2: Comparison: Placebo vs TAK-861 2 mg and 5 mg; Test type: Superiority; p = 0.216, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; LS Mean Difference Estimate = -3.06, 95% CI 2-sided [-6.18 to 0.06], Standard Error of Mean 1.59

3. Secondary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not the occurrence is considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE whose date of onset occurred on or after the first dose of study drug.
Time Frame: From first dose of the study drug up to end of the study (up to 3 months)
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg
Number analyzed (Participants) | 24 | 23 | 24
Participants | 8 | 10 | 18

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to end of the study (up to 3 months)
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo tablets (]matching TAK-861, orally, twice daily (BID), from Days 1 to 56.
Arm/Group | Placebo | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 7/23 | 14/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=24) | TAK-861 2 mg BID (N=23) | TAK-861 2 mg and 5 mg (N=24)
Headache (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 2 | 5
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 3 | 8
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT05687916/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT05687916/SAP_001.pdf